CLINICAL TRIAL: NCT05977725
Title: Hemodynamic Assessment of the Hand Arterial Perfusion Through the Ultrasound-Doppler Hand Acceleration Time (HAT) Technique: A Descriptive Study
Brief Title: Hand Acceleration Time Assessment With Ultrasound Doppler
Acronym: HAT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitari de Bellvitge (Other)
Responsible Party: Principal Investigator, Begoña Gonzalo Villanueva, Expert Vascular Surgeon, Hospital Universitari de Bellvitge
Other Study IDs: 1 - VASC - 2023
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Upper Limb Ischemia; Vascular Disease
Keywords: Hand acceleration time; Upper limb ischemia; Vascular disease
MeSH Terms: conditions — Vascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Lack of upper limb arterial disease.
  Interventions: Diagnostic Test: Hand Doppler Ultrasound
- Patients with Chronic Upper Limb Ischemia: Known diagnosis of chronic upper limb ischemia.
  Interventions: Diagnostic Test: Hand Doppler Ultrasound

INTERVENTIONS:
Diagnostic Test: Hand Doppler Ultrasound — Hand Doppler Ultrasound to assess the Hand Acceleration Time (HAT)

SUMMARY:
Chronic upper limb ischemia syndrome is uncommon compared to lower limb ischemia, with several potential causes (e.g., arteriosclerosis, compressive syndromes, arteritis, connective tissue diseases, trauma, and thrombosis). Many patients with upper limb ischemia remain asymptomatic due to arterial collateral vascularization.

Given the wide variety of potential causes for upper limb ischemia, the diagnosis may require different technical approaches. Doppler ultrasound is a non-invasive, accessible, non-radiating technique that provides direct arterial imaging, yielding valuable information on arterial anatomy and hemodynamics.

Some authors have described the reliability of the arterial duplex ultrasound for lower limb assessment using the pedal acceleration time (PAT). The PAT provides real-time hemodynamic physiological information on the entire limb. The acceleration time (AT) is an ultrasound parameter which measures the time elapsed (in milliseconds, ms) from the beginning of the arterial Doppler waveform until the systolic peak, evaluating the morphology of the arterial waveform in real time. In a healthy individual, this time should be short (between 40 - 100 milliseconds), displaying a triphasic waveform with a systolic acceleration, a sudden diastolic fall, and a subsequent anterograde flow at the end of diastole. A more damped wave suggests proximal stenosis and the acceleration time has been correlated to different degrees of foot ischemia.

Notably, the AT parameter has also been studied in other territories, such as the carotid and pulmonary arteries, coronary arteries, and the aorta. Hand acceleration time (HAT) has also been described very recently as a potential tool to assess hemodialysis access-induced ischemia, cardiogenic shock, and subclavian iatrogenic ischemic lesion. However, the HAT has not yet been properly characterized or validated. Our working hypothesis is that the HAT is a useful diagnostic tool for chronic upper limb ischemia.

ELIGIBILITY:
Inclusion Criteria (healthy volunteers):

* Healthy adult volunteers (≥ 18 years of age).
* No evidence of upper limb arterial disease.
* Who sign the written informed consent.

Exclusion Criteria (healthy volunteers):

* Healthy volunteers unable (at the investigator discretion) to understand or comply with any study-related procedure.
* Healthy volunteers who refuse to participate.
* Those presenting cardiovascular risk factors (e.g., hypertension, diabetes mellitus, dyslipidemia).

Inclusion Criteria (upper limb ischemia patients):

* Adult patients (≥ 18 years of age) with a known diagnosis of chronic upper limb ischemia.
* Who sign the written informed consent.

Exclusion Criteria (upper limb ischemia patients):

* Patients unable (at the investigator discretion) to understand or comply with any study-related procedure.
* Patients who refuse to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of healthy volunteers accompanying patients to the Angiology and Vascular Surgery outpatient clinic visit and patients diagnosed with chronic upper limb ischemia. Both will be required to sign the written informed consent before joining the study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Median (range) hand acceleration time measured by Doppler ultrasound | Day 1
  The hand acceleration time will be measured at the following arteries:
  * Distal radial artery
  * Distal ulnar artery
  * Princeps pollicis artery
  * Index finger radial artery
  * Second common palmar digital artery
  * Fourth common palmar digital artery

SECONDARY OUTCOMES:
Median (range) age of the participants. | Day 1
Number (percentage) of male/female participants. | Day 1
Number (percentage) of patients presenting cardiovascular risk factors of interest. | Day 1
  Cardiovascular risk factors of interest are smoking habits, arterial hypertension, diabetes mellitus, and dyslipidemia).
Number (percentage) of patients with past medical history of interest. | Day 1
  A past medical history of interest is defined as ischemic cardiopathy, heart failure, and chronic obstructive pulmonary disease.
Presence (Yes/No) of distal pulses in the upper limb. | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Background] Sommerset J, Karmy-Jones R, Dally M, Feliciano B, Vea Y, Teso D. Plantar Acceleration Time: A Novel Technique to Evaluate Arterial Flow to the Foot. Ann Vasc Surg. 2019 Oct;60:308-314. doi: 10.1016/j.avsg.2019.03.002. Epub 2019 May 8. PMID 31075481
- [Background] Teso D, Sommerset J, Dally M, Feliciano B, Vea Y, Jones RK. Pedal Acceleration Time (PAT): A Novel Predictor of Limb Salvage. Ann Vasc Surg. 2021 Aug;75:189-193. doi: 10.1016/j.avsg.2021.02.038. Epub 2021 Apr 3. PMID 33823258
- [Background] Strosberg DS, Haurani MJ, Satiani B, Go MR. Common carotid artery end-diastolic velocity and acceleration time can predict degree of internal carotid artery stenosis. J Vasc Surg. 2017 Jul;66(1):226-231. doi: 10.1016/j.jvs.2017.01.041. Epub 2017 Apr 5. PMID 28390773
- [Background] Wang S, Wang Y, Gao M, Tan Y. Acceleration time to Ejection time ratio in fetal pulmonary artery system can predict neonatal respiratory disorders in gestational diabetic mellitus women. Clin Hemorheol Microcirc. 2022;80(4):497-507. doi: 10.3233/CH-211265. PMID 34924370
- [Background] Takemoto K, Hirata K, Wada N, Shiono Y, Komukai K, Tanimoto T, Ino Y, Kitabata H, Takarada S, Nakamura N, Kubo T, Tanaka A, Imanishi T, Akasaka T. Acceleration time of systolic coronary flow velocity to diagnose coronary stenosis in patients with microvascular dysfunction. J Am Soc Echocardiogr. 2014 Feb;27(2):200-7. doi: 10.1016/j.echo.2013.10.013. Epub 2013 Dec 15. PMID 24345631
- [Background] Zarzecki MP, Popieluszko P, Zayachkowski A, Pekala PA, Henry BM, Tomaszewski KA. The surgical anatomy of the superficial and deep palmar arches: A Meta-analysis. J Plast Reconstr Aesthet Surg. 2018 Nov;71(11):1577-1592. doi: 10.1016/j.bjps.2018.08.014. Epub 2018 Aug 24. PMID 30245020
- [Derived] Gonzalo B, Videla S, Moranas J, Carnaval T, Herranz C, Espinar E, Iborra E. Hemodynamic Assessment of Arterial Perfusion by Using the Ultrasonographic Hand Acceleration Time: Protocol for a Cross-Sectional Prospective Descriptive Study. JMIR Res Protoc. 2025 Aug 21;14:e64450. doi: 10.2196/64450. PMID 40839871